CLINICAL TRIAL: NCT04656054
Title: Comparing the Changes in Hemoglobin Level, Coagulopathy Profile and Electrolyte Balance in Large Volume Liposuction Patients But in Different Surface Areas.
Brief Title: Hemoglobin Level, Coagulopathy Profile and Electrolyte Balance
Status: Completed | Type: Observational
Sponsor: Alaa Hassan M. Elhawary (Other)
Responsible Party: Sponsor-Investigator, Alaa Hassan M. Elhawary, Residant doctor at plastic surgery department, Assiut University hospital., Assiut University
Organization: Assiut University (Other)
Other Study IDs: large volume liposuction
Record Dates: First submitted 2020-04-05; First posted 2020-12-07 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2024-02

CONDITIONS: Lipodystrophy; Obesity
Keywords: Liposuction.; Large volume.; electrolyte imbalance.
MeSH Terms: conditions — Lipodystrophy; Obesity | interventions — Lipectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: liposuction — liposuction procedure and observation of the hematological changes on the patients

SUMMARY:
What is Impact of Amount Versus Surface Area of Liposuction on Haematological Parameters, Coagulopathy Profile and Electrolyte Balance? Liposuction involves the creation of extensive subsurface trauma, comparable in many respects to the massive injury of an internal burn. Liposuction commences with cannula aspiration of several liters of fluid-engorged adipose tissue, during which small feeder vessels are inevitably torn.

Operating on multiple areas increases the area of injury regardless of whether just small amounts of fat are removed. Because many of the complications associated with large volume liposuction are related to fluid shifts and fluid balance, classifying the procedure based on the total volume removed from the patient, including fat, wetting solution, and blood, makes more sense to evaluate the damage made by the procedure.

Safety and aesthetic issues define large-volume liposuction as having a 5,000-ml aspirate, mega-volume liposuction as having an 8,000-ml aspirate, and giganto-volume liposuction as having an aspirate of 12,000 ml or more.

DETAILED DESCRIPTION:
Liposuction is fat- removing aesthetic surgery procedure that aims to body contouring. Liposuction is the most frequently performed aesthetic surgery procedure in Western Countries. This technique has had rapid development since the 1970s, when it was experimented for the first time by A. and G. Fischer. It is currently widely used in clinical practice for many different situations in aesthetic, reconstructive and functional fields.

At 1970s, fat removal was carried out with a blunt curette. This technique was modified in 1977 by a French surgeon, Yves Gerard Illouz, who added hyaluronidase and saline to emulsify the fatty tissue, and hence facilitate aspiration with the use of liposuction cannula. This was termed the 'wet technique' and was introduced to reduce blood loss during the procedure.

The current options for wetting solutions are dry, wet, superwet, and tumescent. The dry technique employs no wetting solution and has few indications in liposuction. The wet technique involves instillation of 200 to 300 mL of solution per area to be treated, regardless of the amount aspirated. The superwet technique employs an infiltration of 1 mL per estimated mL of expected aspirate, and this is the technique practiced at our institution. Tumescent infiltration, popularized by Klein, involves infiltration of wetting solution that creates significant tissue turgor and results in infiltration of 3 to 4 mL of wetting solution per mL aspirated. Regardless of technique, the infiltrate should be allowed to take effect for seven minutes prior to suctioning.

Most studies consider the most important parameter, to determine the safety of liposuction, is the amount (volume) of aspirated fluid. A review of the scientific literature shows that there are no scientific data available to support a specific volume maximum at which point liposuction is no longer safe, although the risk of complications is unavoidably higher as the volume of aspirate and the number of anatomic sites treated increase.

Safety and aesthetic issues define large-volume liposuction as having a 5,000-ml aspirate, mega-volume liposuction as having an 8,000-ml aspirate, and giganto-volume liposuction as having an aspirate of 12,000 ml or more.

In large volume liposuction, there is potential for large fluid shifts secondary to the volume of tissue removed, with a risk of developing pulmonary edema, high-volume liposuction is significantly more prone to complications than the original form of liposuction.

There is a long history of debate over the safe volume of fat tissue that can be removed by liposuction. Current ASPS guidelines define 5,000 milliliters (five liters) as "large-volume liposuction" potentially associated with a higher risk of complications. But the guidelines acknowledge there is no scientific data to support an absolute cutoff point. Patients with complications had larger liposuction volumes-average 3.4 liters-and higher BMIs. Patients undergoing "large-volume" liposuction of more than five liters had a higher overall complication rate: 3.7 versus 1.1 percent.

On the other hand, liposuction involves the creation of extensive subsurface trauma, comparable in many respects to the massive injury of an internal burn. Liposuction commences with cannula aspiration of several liters of fluid-engorged adipose tissue, during which small feeder vessels are inevitably torn.

Only few studies have mentioned the effect of surface area on liposuction and none of those studies have been published at certified impacted magazine.

In this study considers the amount of liposuction is a constant factor (Large volume liposuction) and the surface area is the variant to detect the changes in hemogram, coagulation profile and electrolyte imbalance that may lead to possible complication.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient.
2. Age: 25-45 years.
3. BMI <40
4. Large volume liposuction
5. Patient asking for liposuction or suction assisted lipoectomy.

Exclusion Criteria:

1. Male patient.
2. Age >45 or <25 years.
3. Uncontrolled chronic diseases as DM, HTN.
4. Show degrees of lipodystropy at breast.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: To assess the impact of amount, up to 8 litres, versus surface area of liposuction on haematological parameters, coagulopathy profile and electrolyte balance.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Comparing the blood hemoglobin level pre, intra and post operative between two groups of patients, both have done large volume liposuction, with different surface areas liposuctioned. | 1 year
  To compare the impact of large volume liposuction (5 to 8 liters) from different body surface areas on the patient's hemoglobin level preoperatively, intraoperative and postoperatively.
  The surface area will be calculated according to Lund and Browder chart by percentage (the most accurate and widely used chart to calculate total body surface area affected by a burn injury) The volume is measured by Liters. Hemoglobin level is measured by g/dl.
Comparing the coagulation profile (mainly prothrombin concentration and INR) pre, intra and post operative between two groups of patients, both have done large volume liposuction, with different surface areas liposuctioned. | 1 year
  To compare the impact of large volume liposuction (5 to 8 liters) from different body surface areas on the patient's Coagulopathy Profile (prothrombin concentration, INR) preoperatively, intraoperative and postoperatively.
  The surface area will be calculated according to Lund and Browder chart by percentage (the most accurate and widely used chart to calculate total body surface area affected by a burn injury) The volume is measured by Liters. The coagulation profile includes mainly prothromin concentration( measured by percentage) and INR.
Comparing potassium serum ions level pre, intra and post operative between two groups of patients, both have done large volume liposuction, with different surface areas liposuctioned. | 1 year
  To compare the impact of large volume liposuction (5 to 8 liters) from different body surface areas on the patient's electrolyte balance preoperatively, intraoperative and postoperatively.
  The surface area will be calculated according to Lund and Browder chart by percentage (the most accurate and widely used chart to calculate total body surface area affected by a burn injury)
  The volume is measured by Liters.
  The electrolyte, that are included in the study, is potassium ions measured by mmol/L.
Comparing the blood hematocrit level pre, intra and post operative between two groups of patients, both have done large volume liposuction, with different surface areas liposuctioned. | 1 year.
  To compare the impact of large volume liposuction (5 to 8 liters) from different body surface areas on the patient's hemoglobin level preoperatively, intraoperative and postoperatively.
  The surface area will be calculated according to Lund and Browder chart by percentage (the most accurate and widely used chart to calculate total body surface area affected by a burn injury) The volume is measured by Liters. Hematocrit level is measured by percentage.
Comparing the sodium serum ions level pre, intra and post operative between two groups of patients, both have done large volume liposuction, with different surface areas liposuctioned. | 1 year.
  To compare the impact of large volume liposuction (5 to 8 liters) from different body surface areas on the patient's electrolyte balance preoperatively, intraoperative and postoperatively.
  The surface area will be calculated according to Lund and Browder chart by percentage (the most accurate and widely used chart to calculate total body surface area affected by a burn injury)
  The volume is measured by Liters.
  The electrolyte, that are included in the study, is sodium ions measured by mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Assem H. Abdelhafez, professor, Study Chair — Assiut University
Locations (1):
- Assuit University, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No